CLINICAL TRIAL: NCT01509404
Title: Cytogam Administration in Abdominal Organ Transplant Recipients at High Risk for CMV Infection
Brief Title: Cytogam Administration in Abdominal Organ Transplant Recipients at High Risk for Cytomegalovirus Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00009601
Record Dates: First submitted 2012-01-10; First posted 2012-01-13 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Cytomegalovirus Disease
Keywords: CMV; cytomegalovirus; transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir; cytomegalovirus-specific hyperimmune globulin

ARMS (2):
- Valcyte (Active Comparator): valganciclovir per package insert guidelines for prophylaxis against CMV infection for 200 days post-transplant
  Interventions: Drug: Valganciclovir
- Valcyte then Cytogam (Active Comparator): valganciclovir per package insert guidelines for 100 days post-transplant with Cytogam 100 mg/kg administered at 90 days, 120 days, and 180 days post-transplant for prophylaxis against CMV infection
  Interventions: Biological: CMV hyperimmune globulin; Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Valcyte per package insert guidelines for 200 days post transplant
  Other Names: Valcyte
  Arms: Valcyte
Biological: CMV hyperimmune globulin — 100 mg/kg administered at 90 days, 120 days, and 180 days post-transplant
  Other Names: Cytogam
  Arms: Valcyte then Cytogam
Drug: Valganciclovir — valganciclovir per package insert guidelines for prophylaxis against CMV infection for 200 days post-transplant
  Other Names: Valcyte
  Arms: Valcyte then Cytogam

SUMMARY:
The purpose of the study is to assess the incidence and severity of late Cytomegalovirus (CMV) disease, defined as CMV syndrome or tissue invasive disease occurring between 100 and 200 days and after 200 days post-transplant in patients treated with valganciclovir per package insert guidelines for prophylaxis against CMV infection for 200 days post-transplant versus valganciclovir per package insert guidelines for 100 days post-transplant with Cytogam 100 mg/kg administered at 90 days, 120 days, and 180 days post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years of age.
2. Male or female patients who CMV seronegative receiving a kidney, pancreas or liver from a seropositive donor.
3. Female patients of child bearing potential must have a negative urine or serum pregnancy test within the past 48 hours prior to receiving transplant or study inclusion.
4. The patient has given written informed consent to participate in the study.

Exclusion Criteria:

1. Solid organ transplant recipient is CMV seropositive at the time of transplant.
2. Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV).
3. Patient has uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives.
4. Patients with thrombocytopenia (<25,000/mm3 ), with an absolute neutrophil count of < 1,000/mm3); and/or leucopoenia (< 2,000/mm3), or anemia (hemoglobin < 6 g/dL) prior to study inclusion.
5. Patient is taking or has been taking an investigational drug in the 30 days prior to transplant.
6. Patient has a known hypersensitivity to valganciclovir, tacrolimus, mycophenolate mofetil, rabbit anti-thymocyte globulin, CMV hyperimmune globulin, basiliximab or corticosteroids.
7. Patients with severe diarrhea or other gastrointestinal disorders that might interfere with their ability to absorb oral medication.
8. Patient is pregnant or lactating, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive human Chorionic Gonadotropin (hCG) laboratory test.
9. Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.
10. Inability to cooperate or communicate with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valcyte | Valcyte Then Cytogam
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Valcyte - Kidney Transplant: Subjects who received a kidney transplant and assigned to the Valcyte only Treatment arm.
- Valcyte Then Cytogam - Kidney Transplant: Subjects who received a kidney transplant and assigned to the Valcyte then CytogamTreatment arm.
- Valcyte - Liver Transplant: Subjects who received a liver transplant and assigned to the Valcyte only Treatment arm.
- Valcyte Then Cytogam - Liver Transplant: Subjects who received a liver transplant and assigned to the Valcyte then Cytogam Treatment arm.
- Total: Total of all reporting groups
Arm/Group | Valcyte - Kidney Transplant | Valcyte Then Cytogam - Kidney Transplant | Valcyte - Liver Transplant | Valcyte Then Cytogam - Liver Transplant | Total
Number analyzed (Participants) | 17 | 15 | 3 | 5 | 40
Age, Continuous [Mean (Full Range); unit: years] | 51 [21 to 71] | 54 [26 to 69] | 58 [27 to 58] | 60 [48 to 61] | 56 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 0 | 10
  Male | 13 | 11 | 1 | 5 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 0 | 0 | 13
  White | 9 | 9 | 3 | 5 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Retransplant [Count of Participants; unit: Participants] | 2 | 2 | 0 | 0 | 4
Weight (kg) [Mean (Standard Deviation); unit: kg] | 71 (20) | 88 (21) | 84 (13) | 91 (25) | 84 (20)
Pre-emptive [Count of Participants; unit: Participants] — Population: Pre-Emptive applies only to kidney transplant patients. Pre-emptive values were obtained by counting the number of patients who were not on dialysis prior to their kidney transplant.
  Participants
    number analyzed (Participants) | 17 | 15 | 0 | 0 | 32
    (all) | 3 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Late CMV Disease
Description: Number of any clinically significant late CMV disease, defined as CMV syndrome or tissue-invasive disease occurring after the first 200 days post transplant
Time Frame: after 200 days post-transplant until 2 years post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0

2. Secondary Outcome: Number of Patients With Early CMV Infection
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
Participants | 3 | 1

3. Secondary Outcome: Number of Patients With Cell Mediated Immunity
Description: Positive CMV quantiferon at last follow-up
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
Participants | 8 | 13

4. Secondary Outcome: Renal Function
Description: Renal function will be assessed by an estimated creatinine clearance utilizing the abbreviated Modification of Diet in Renal Disease (MDRD) equation at 6, 12, and 24 months after transplant
Time Frame: 6, 12, and 24 months after transplant
Measure: Mean (Full Range); unit: mL/min/1.73m^2
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
mL/min/1.73m^2
  GFR at 180 Days | 57 [22 to 123] | 53 [30 to 78]
  GFR at 1 year | 59 [26 to 171] | 54 [31 to 71]
  GFR at 2 years | 59 [29 to 143] | 55 [20 to 72]

5. Secondary Outcome: Number of Participants With Acute Cellular and/or Antibody Mediated Rejection
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
Participants | 2 | 6

6. Secondary Outcome: Number of Participants With Opportunistic Infections
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
Participants | 17 | 19

7. Secondary Outcome: Number of Participants With Asymptomatic CMV Viremia
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
Participants | 1 | 5

8. Secondary Outcome: Number of Participants With CMV Seroconversions
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Valcyte | Valcyte Then Cytogam
Number analyzed (Participants) | 20 | 20
Participants | 13 | 19

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Valcyte | Valcyte Then Cytogam
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20 | 4/20
Other Adverse Events (participants affected / at risk) | 16/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valcyte (N=20) | Valcyte Then Cytogam (N=20)
CMV disease (Infections and infestations) | 3 (3) | 4 (4)
Graft loss (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valcyte (N=20) | Valcyte Then Cytogam (N=20)
Leukopenia (Blood and lymphatic system disorders) | 9 (9) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
BK infection (Renal and urinary disorders) | 3 (3) | 5 (5)
Candidiasis (Infections and infestations) | 0 (0) | 3 (3)
Acute rejection (Renal and urinary disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No